CLINICAL TRIAL: NCT05463419
Title: A Phase II/III, Randomized, Double-blinded Study to Evaluate the Efficacy, Safety and Immunogenicity of a Booster Dose of PIKA Recombinant SARS-CoV-2 Vaccine in Adults Who Received 2 or More Doses of Inactivated Covid-19 Vaccine.
Brief Title: A Phase II/III Study of PIKA Recombinant SARS-CoV-2 Vaccine as a Booster Dose.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: YS302
Record Dates: First submitted 2022-06-29; First posted 2022-07-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-10

CONDITIONS: Covid-19 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIKA COVID-19 vaccine (Experimental): One dose of the experimental vaccine should be administered on Study Day 0 in the deltoid muscle.
  Interventions: Biological: PIKA COVID-19 vaccine
- Inactivated Covid-19 vaccine (Active Comparator): One dose of the control vaccine should be administered on Study Day 0 in the deltoid muscle.
  Interventions: Biological: Inactivated Covid-19 vaccine

INTERVENTIONS:
Biological: PIKA COVID-19 vaccine — SARS-CoV-2 spike subunit protein (Also called "Recombinant SARS-CoV-2 S-trimer protein"), PIKA adjuvant.
  Arms: PIKA COVID-19 vaccine
Biological: Inactivated Covid-19 vaccine — Inactivated SARS-CoV-2 virus
  Arms: Inactivated Covid-19 vaccine

SUMMARY:
This is a Phase II/III, randomized, double-blinded study in adults ≥ 18 years old who received 2 or more doses of inactivated COVID-19 vaccine to evaluate the efficacy, safety and immunogenicity of a booster dose of PIKA COVID-19 vaccine compared to the comparator inactivated COVID-19 vaccine. Phase II/III will be a competitive enrollment process in all participating countries. Once the target number of subjects is reached, the enrollment in all participating countries in the particular phase will be stopped.

DETAILED DESCRIPTION:
In phase II, a total of 300 eligible subjects will be randomly allocated in a 1:1 ratio to receive PIKA COVID-19 vaccine or the comparator inactivated COVID-19 vaccine. The ratio of the GMT of neutralizing antibody on Day 14 after the booster dose of PIKA COVID-19 vaccine group and inactivated COVID-19 vaccine group will be calculated. Based on the Phase I immunogenicity data of PIKA vaccine, the proposed Phase II sample size results in nearly 100% power in a two-sample t test of the log- transformed neutralizing antibody titers with a two-sided alpha=0.05. Among 300 subjects, at least 200 subjects will be enrolled as subset of long term immunogenicity and 100 subjects will be enrolled as subset of early immunogenicity. Among the 100 early immunogenicity subset, the ratio of the GMT of neutralizing antibody on Day 7 after the booster dose of PIKA COVID-19 vaccine group and inactivated COVID-19 vaccine group will be calculated. Therefore, the 100 subjects randomized to the early immunogenicity subset will have additional blood sampling on Day 7. After completion of the 7-day safety observation following the immunization of all subjects in the Phase II trial, a Safety Monitoring Committee (SMC) meeting will be held to determine whether to initiate enrollment of participants in the Phase III trial. In phase III, total 9,000 eligible subjects will be randomly allocated in a 1:1 ratio to the PIKA COVID-19 vaccine group or the comparator inactivated COVID-19 vaccine group. The sample size provides an approximately 90% power to detect a protection rate of at least 65% by PIKA vaccine in a Poisson regression analysis with a one-sided alpha of 0.025. The calculations consider an interim analysis performed with 50% of the information collected using a Pocock boundary to adjust for multiplicity. A 1% infection rate in the control group and an approximately a 10% attrition rate are assumed. It is of note that while the actual background incidence rate can vary, the sample size requirement amounts to achieving an observation of 82 COVID-19 cases to ensure the statistical power under the 65% protection rate assumption. Similarly, the interim analysis will need to be conducted at when approximately 41 cases are observed to maintain the planned operating characteristics. Among total subjects, at least 6% subjects will be enrolled as subset of immunogenicity. Eligible subjects will receive a dose of investigational vaccine via intramuscular injection in deltoid muscle on Day 0. All subjects will be monitored for at least 30 minutes after injection. Solicited AEs will be recorded for 7 days. Unsolicited AEs and MAAEs will be recorded for 28 days following injection. SAEs, SUSARs, AESIs will be recorded for the entire duration of the study. It will take about 13 months for each subject from enrollment to the last visit. Some subjects may withdraw or discontinue from the study during the study for any reason.

ELIGIBILITY:
Inclusion Criteria:

Subject who met all of the following criteria may be enrolled.

1. Age more than or equal 18 years on Screening.
2. Judged by the investigator to be healthy based on medical history, physical examination and vital signs performed at screening.
3. Able to provide informed consent.
4. Able and willing to comply with all study procedures over follow up period of approximately 12 months.
5. Received 2 or more doses of inactivated COVID-19 vaccine as primary series with their last dose at least 3 months prior to enrollment.
6. Axillary body temperature ≤37.5℃.
7. SARS-COV-2 test was negative for nasopharyngeal swabs by RT PCR.
8. Non-pregnant and not lactating women.
9. For female subjects of childbearing potential: must agree to avoid pregnancy from Study Day 0 to Study Day 60 during the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide.
10. Male subjects who are sexually active with a woman of childbearing potential and have not had vasectomy must agree to practice a highly effective form of contraception with their female partners of childbearing potential during the trial, starting after screening until 60 days after receiving the last vaccination.
11. Men must be willing to refrain from sperm donation, starting after screening until 60 days after receiving the last vaccination.

Exclusion Criteria:

* Subject who met any of the following criteria may not be enrolled.

  1. Abnormal vital signs or laboratory test results prior to D0 judged as clinically significant by investigator.
  2. Known allergy, hypersensitivity, or intolerance to the test vaccine (including any excipients and the antibiotics kanamycin and aminoglycosides).
  3. History of severe allergies to any drugs, foods or vaccines, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.
  4. Diagnosed with any serious disease, or congenital malformation, or uncontrolled chronic disease that may influence the compliance with the study including but not limited to respiratory disease such as asthma or chronic bronchitis, serious cardiovascular disease, kidney disease, autoimmune disease, thalassemia, malignant tumor, hereditary allergy, etc.
  5. History or family history of convulsions, seizures, encephalopathy, and mental illness.
  6. History of narcolepsy.
  7. Known substance abuse and addiction within the past 2 years.
  8. Uninterrupted use of systemic immunosuppressants or other immunomodulators within 30 days prior to D0.
  9. Use of blood or blood-related products (e.g., blood transfusion, human albumin, human immunoglobulin, etc.) within 30 days prior to D0.
  10. Blood loss >400 mL within 28 days prior to D0 (e.g., donated blood or blood products or injury), or planned to donate blood or plasma before D28 of the study.
  11. Use of nonsteroidal anti-inflammatory drugs and/or antiallergic drugs within 3 days prior to D0
  12. Have symptoms of COVID-19, such as respiratory symptoms, fever, cough, shortness of breath and dyspnea.
  13. Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating IM vaccination based on Investigator's judgment.
  14. Surgical removal of whole or part of spleen for any reason
  15. Received any vaccines within 28 days prior to D0 or disagree to avoid receiving any vaccines before D28 of the study except the emergent vaccination such as rabies vaccine, tetanus vaccine.
  16. Participating in or planning to participate in other clinical trials (drugs or vaccines) during the study period.
  17. Any other conditions not eligible for participating in the study at investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5860 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Immunogenicity at Phase II Study | at day 14 after booster.
  Geometric mean titer (GMT) of neutralizing antibody against Omicron virus on D14 after the booster dose
Efficacy at Phase III Study | up to 360 days after booster
  Incidence of first occurrence of Rt-PCR positive symptomatic illness after D14 of booster dose
Safety at Phase II and Phase III | up to 360 days after booster.
  Incidence of AE, MAAE, SAE, SUSAR and AESI after booster dose

SECONDARY OUTCOMES:
Immunogenicity at Phase II Study | at day 7, day 14, day 90, day 180, day 360 after booster.
  GMT of neutralizing antibody against wild type SARS-CoV-2 virus on Day 7, Day 14, Day 90, Day 180, Day 360.
  * GMT of neutralizing antibody against Omicron virus on Day 7.
  * Seroconversion rate of neutralizing antibody against wild type SARS-CoV-2 virus from Day 0 to Day 7.
  * Seroconversion rate of neutralizing antibody against Omicron virus from Day 0 to Day 7.
  * Mean geometric titers fold growth of neutralizing antibody against wild type SARS-CoV-2 virus from Day 0 to Day 7.
  * Mean geometric titers fold growth of neutralizing antibody against Omicron virus from Day 0 to Day 7.
  * GMT of serum IgG antibody on Day 7.
  * Seroconversion rate of serum IgG antibody from Day 0 to Day 7.
Efficacy at Phase III Study | from day 14 to day 360 after booster.
  Incidence of the first occurrence of either COVID-19 or SARS CoV-2 infection regardless of symptomatology or severity starting 14 days after the booster dose.
  For immunogenicity subset (6% of Phase III):
  * GMT of neutralizing antibody against Omicron virus on Day 7 and Day 14.
  * Seroconversion rate of neutralizing antibody against Omicron virus from Day 0 to Day 7 and Day 14.
  * Mean geometric titersfold growth of neutralizing antibody against Omicron virus from Day 0 to Day 7 and Day 14.
  * GMT of serum IgG antibody on Day 7 and Day 14.
  * Seroconversion rate of serum IgG antibody from Day 0 to Day 7, Day 14

CONTACTS AND LOCATIONS:
Locations (6):
- Philippines (5):
  - Health Index Multispecialty Clinic -Clinical Research, Cavite
  - Norzel Medical and Diagnostic Clinical, Cebu
  - Tropical Disease Foundation, City of Muntinlupa
  - St. John Hospital, Naga
  - UERM Research Center, Quezon City
- Al Kuwait Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim RJ, Qiu X, Alberto E, Capeding MR, Carlos J, Leong RN, Gutierrez JL, Trillana M, Liu Y, Mojares Z. Safety and immunogenicity of PIKA-adjuvanted recombinant SARS-CoV-2 spike protein subunit vaccine as a booster against SARS-CoV-2: a phase II, open-label, randomized, double-blinded study. Clin Exp Vaccine Res. 2024 Oct;13(4):329-337. doi: 10.7774/cevr.2024.13.4.329. Epub 2024 Oct 31. PMID 39525672